CLINICAL TRIAL: NCT01179490
Title: A Multicenter, Open-Label, Phase 2 Study of SyB L-0501 (Bendamustine Hydrochloride) for Patients With Multiple Myeloma
Brief Title: Efficacy and Safety Study of SyB L-0501 for Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010002
Record Dates: First submitted 2010-08-02; First posted 2010-08-11 (Estimated); Results first posted 2013-03-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SyB L-0501 + prednisolone (Experimental): SyB L-0501 (150 mg/m2/day) will be administered by intravenous drip infusion for 60 min for 2 consecutive days and the course will be observed for the next 26 days. This is taken as one cycle and administration is repeated for 2-9 cycles (when a plateau is not reached after nine cycles, administration of up to an additional three cycles for a maximum of 12 cycles is possible. Prednisolone (60 mg/m2/day) will be administered orally for 4 consecutive days and the course will be observed for the next 24 days.
  Interventions: Drug: SyB L-0501; Drug: prednisolone

INTERVENTIONS:
Drug: SyB L-0501 — SyB L-0501 (150 mg/m2/day) will be administered by intravenous drip infusion for 60 min for 2 consecutive days and the course will be observed for the next 26 days. This is taken as one cycle and administration is repeated for 2-9 cycles (when a plateau is not reached after nine cycles, administration of up to an additional three cycles for a maximum of 12 cycles is possible).
Drug: prednisolone — Prednisolone will be administered (60 mg/m2/day) orally for 4 consecutive days and the course will be observed for the next 24 days.

SUMMARY:
The study objectives of this study are to determine the effects, safety, and pharmacokinetics of bendamustine for multiple myeloma to a regimen of bendamustine and prednisolone.

DETAILED DESCRIPTION:
The study objectives of this study are to determine the effects, safety, and pharmacokinetics of bendamustine for untreated and maladjustment to hematopoietic stem cell transplantation (HSCT) multiple myeloma to a regimen of bendamustine and prednisolone.

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if all of the following criteria are met: Patients confirmed to have multiple myeloma (symptomatic myeloma) defined in the diagnostic criteria of the International Myeloma Working Group (IMWG).

* Patients with measurable lesions
* Patients with no history of treatment (no history of chemotherapy or radiotherapy)
* Patients should not be considered candidates for high dose therapy/autologous stem cell transplantation due to coexistent medical conditions, advanced age, poor performance status, refusal of high dose chemotherapy, or other reasons as judged by the patient and/or physician.
* Expected survival of at least 3 months
* Patients aged between 20 and 79 years (at the time of provisional registration)
* Performance status (P.S.) grade 0-2. P.S. 3 possible only for osteolytic lesions
* Patients with adequately maintained organ function (e.g., bone marrow, heart, lungs, liver, kidneys,)
* Patients from whom written consent to participate in this study has been obtained.

Exclusion Criteria:

Patients are excluded from participating in the study if 1 or more of the following criteria are met:

* Patients with apparent infections (including viral infections)
* Patients with serious complications (hepatic failure, renal failure, or diabetes with insulin administration)
* Patients with complications or a medical history of serious cardiac disease (e.g., myocardial infarction, ischemic heart disease) within 2 years before preliminary registration. Patients with arrhythmia requiring treatment.
* Patients with serious gastrointestinal symptoms (profound or serious nausea / vomiting or diarrhea, etc.)
* Patients who were hepatitis B virus antigen (HBsAG)-positive, hepatitis C virus (HCV) antibody-positive or human immunodeficiency virus (HIV) antibody-positive
* Patients with a serious bleeding tendency [e.g., Disseminated intravascular coagulation (DIC)]
* Patients with interstitial pneumonia, pulmonary fibrosis or pulmonary emphysema requiring treatment, or such diseases in the past
* Patients with apparent amyloidosis as a complication
* Patients with clinical symptoms of invasion or suspected invasion of the central nervous system.
* Patients with active multiple cancers
* Patients who have or previously had autoimmune hemolytic anemia.
* Patients administered this investigational drug in the past
* Patients who received hematopoietic stem cell transplantation in the past.
* Patients who received cytokines such as granulocyte colony stimulating factor (G-CSF) or erythropoietin or a blood transfusion within 1 week before the screening examination prior to preliminary registration for this study
* Patients who were administered an investigational drug during a clinical study or an unapproved drug within 3 months prior to preliminary registration in this study
* Patients with prior allergies to medications similar to the investigational drug (e.g., alkylating agents, or purine nucleotide analogs), mannitol or prednisolone
* Patients with drug addiction, narcotic addiction or alcoholism.
* Patients who were pregnant, breastfeeding women or who had a possibility to be pregnant
* Patients who do not agree to contraception during the following periods. For males, during or for 6 months after completion of administration of the investigational drug. For females, during or for 3 months after completion of administration of the investigational drug
* Patients whom the investigator or the sub-investigators considered to be inappropriate for the study

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shinsuke Iida, MD, Ph D, Study Chair — Nagoya City University Graduate School of Medical Sciences
Locations (3):
- Japan (3):
  - Research site, Nagoya, Aichi-ken
  - Research site, Fukuoka, Fukuoka
  - Research site, Isehara, Kanagawa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SyB L-0501 + Prednisolone
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Age Continuous [Median (Standard Deviation); unit: Year] | 69.0 (2.3)
Age, Customized [Number; unit: Participants]
  20-29 years | 0
  30-39 years | 0
  40-49 years | 0
  50-59 years | 0
  60-69 years | 3
  70-84 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Condition with symptoms of Multiple Myeloma [Number; unit: Participants] — Condition with symptoms of Multiple Myeloma (Development of hyperviscosity syndrome, amyloidosis, Bacterial infection twice or more in a year)
  Participants
    No | 5
    Yes | 0
Previous treatment of multiple myeloma [Number; unit: Participants]
  No | 5
  Yes | 0
Reason for not eligible for hematopoietic stem cell transplantation [Number; unit: Participants]
  Age 66 years or older | 5
  Presence of cardiopulmonary dysfunction | 0
  Renal dysfunction | 0
  Other | 0
Performance status (P.S.) [Number; unit: Participants] — 0: Asymptomatic 1: Symptomatic but completely ambulatory 2: Symptomatic, <50% in bed during the day 3: Symptomatic, >50% in bed, but not bedbound
  Participants
    0 | 3
    1 | 0
    2 | 2
    3 | 0
Clinical stage [International staging system (ISS) category] [Number; unit: Participants] — Stage I: Serum β2-microglobulin (β2M) < 3.5 mg/L and serum albumin ≥ 3.5 g/dL)
  Stage II: Serum β2M ≥3.5 - < 5.5 mg/L; or serum β2M < 3.5 mg/L and serum albumin < 3.5 g/dL)
  Stage III: (Serum β2M ≥ 5.5 mg/L)
  Participants
    Stage I | 0
    Stage II | 3
    Stage III | 2
Previous history of multiple myeloma [Number; unit: Participants]
  No | 5
  Yes | 0
Associated symptom of the primary disease [Number; unit: Participants]
  No | 0
  Yes | 5
Complications of multiple myeloma [Number; unit: Participants]
  No | 0
  Yes | 5
Serum β2M in clinical stage [Median (Standard Deviation); unit: mg/L] | 5.00 (1.48)
Height [Mean (Standard Deviation); unit: cm] | 151.40 (8.53)
Weight [Median (Standard Deviation); unit: kg] | 52.40 (10.41)
Body surface area [Median (Standard Deviation); unit: m2] | 1.470 (0.185)

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate [Based on the Modified Southwest Oncology Group (SWOG) Criteria]
Description: The proportion of subjects evaluated as CR was calculated.
  CR (modified SWOG) requires all of the followings:
  1. Decline in serum myeloma protein by ≥75% to ≤25 g/L
  2. Reduction in 24 h urinary protein by ≥90% to ≤200 mg/24 h
  3. No increase in skeletal destruction
  4. Serum calcium within normal range
  5. No blood transfusion required in the previous 3 months
Time Frame: Up to 36 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Percentage of Participants | 40.0 [5.3 to 85.3]

2. Secondary Outcome: CR Rate [Based on the International Myeloma Working Group (IMWG) Criteria]
Description: The proportion of subjects evaluated as CR [strict CR (sCR) + CR] was calculated.
  sCR (IMWG): CR as defined below plus Normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence
  CR (IMWG): Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow
Time Frame: Up to 36 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Percentage of participants | 0.0 [0.0 to 52.2]

3. Secondary Outcome: Response Rate (Based on the IMWG Criteria)
Description: The proportion of subjects evaluated as response [sCR + CR + very good partial response (VGPR) + Partial Response (PR)] was calculated.
  VGPR (IMWG): Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100mg per 24 h
  PR (IMWG): ≥50% reduction of serum M-protein and reduction in 24 h urinary M-protein by ≥90% or to <200mg per 24 h
Time Frame: Up to 36 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Percentage of participants | 60.0 [14.7 to 94.7]

4. Secondary Outcome: CR Rate Based on the (Bladé) Criteria
Description: The proportion of subjects evaluated as CR was calculated.
  CR (Bladé) requires all of the followings:
  1. Absence of the original monoclonal paraprotein in serum and urine by immunofixation, maintained for a minimum of 6 weeks. The presence of oligoclonal bands consistent with oligoclonal immune reconstitution does not exclude CR.
  2. <5% plasma cells in a bone marrow aspirate and also on trephine bone biopsy, if biopsy is performed. If absence of monoclonal protein is sustained for 6 weeks it is not necessary to repeat the bone marrow, except in patients with non-secretory myeloma where the marrow examination must be repeated after an interval of at least 6 weeks to confirm CR.
  3. No increase in size or number of lytic bone lesions (development of a compression fracture does not exclude response)
  4. Disappearance of soft tissue plasmacytomas
Time Frame: Up to 36 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Percentage of participants | 0.0 [0.0 to 52.2]

5. Secondary Outcome: Response Rate (Based on the Bladé Criteria)
Description: The proportion of subjects evaluated as response (CR + PR) was calculated.
  PR (Bladé) requires 1. or all of the others:
  1. Some, but not all, of the criteria for CR are fulfilled
  2. ≥50% reduction in the level of the serum monoclonal paraprotein, maintained for a minimum of 6 weeks.
  3. Reduction in 24 h urinary light chain excretion either by ≥90% or to <200 mg, maintained for a minimum of 6 weeks.
  4. For patients with non-secretory myeloma only, ≥50% reduction in plasma cells in a bone marrow aspirate and on trephine biopsy, if biopsy is performed, maintained for a minimum of 6 weeks.
  5. ≥50% reduction in the size of soft tissue plasmacytomas (by radiography or clinical examination).
  6. No increase in size or number of lytic bone lesions (development of a compression fracture does not exclude response).
Time Frame: Up to 36 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Percentage of participants | 60.0 [14.7 to 94.7]

6. Secondary Outcome: Response Rate (Based on the Modified SWOG Criteria)
Description: The proportion of subjects evaluated as response (CR + PR) was calculated.
  PR (SWOG) requires the followings:
  1. Decline in myeloma protein of ≥25%-<74% in serum myeloma protein
  2. Reduction in 24h urinary myeloma protein of ≥25%-<89%
  3. No increase in skeletal destruction
  4. Serum calcium within normal range
Time Frame: Up to 36 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Percentage of participants | 60.0 [14.7 to 94.7]

7. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is the period from patient registration to either the date of recurrence, exacerbation, progression or death.
  Recurrence, exacerbation, progression were assessed from serum M-protein, urine M-protein, serum free light chain (FLC), the percentage of marrow plasma cells, disappearance of clonal plasma cells, plasma cell tumor in soft tissue, and bone lesion.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: Days
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Days | 205.0 [38 to 274]

8. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is the period from patient registration to either the date of recurrence, exacerbation, progression, death or discontinuation of treatment.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: Days
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Days | 205.0 [38 to 274]

9. Secondary Outcome: Duration of Response (DOR)
Description: DOR is the period from the date of achieving CR or PR to either the date of recurrence, exacerbation, progression or death.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: Days
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Days | 162.0 [99 to 252]

10. Secondary Outcome: Overall Survival (OS)
Description: OS is the period from the date of patient registration to the date of death.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: Days
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Days | 205.0 [38 to 330]

11. Secondary Outcome: Number of Subjects With Adverse Event, Related Adverse Event, Serious Adverse Event, and Related Serious Adverse Event
Description: Adverse events were evaluated using Common Terminology Criteria for Adverse Events (CTCAE) v4.02, Japan Clinical Oncology Group/Japan Society of Clinical Oncology (JCOG/JSCO) version, and were encoded using Medical Dictionary for Regulatory Activities (MedDRA).
Time Frame: Up to 2 years
Measure: Number; unit: Participants
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Participants
  Subjects with adverse event | 5
  Subjects with related adverse event | 5
  Subjects with serious adverse event | 2
  Subjects with related serious adverse event | 2

12. Secondary Outcome: Number of Adverse Events, Related Adverse Events, Serious Adverse Events, and Related Serious Adverse Events
Description: as for outcome 11
Time Frame: Up to 2 years
Measure: Number; unit: Events
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Events
  Adverse events | 166
  Related adverse events | 155
  Serious adverse events | 4
  Related serious adverse events | 4

13. Secondary Outcome: Number of Subjects With Abnormality (Grade ≥3) in Laboratory Test Values
Description: Abnormalities in laboratory test values in overall study period were analyzed. Severity of abnormalities were evaluated using CTCAE.
  grade 1 : mild
  grade 2 : moderate
  grade 3 : severe or medically significant but not immediately life-threatening
  grade 4 : life threatening or disabling
  grade 5 : death related to AE
Time Frame: Up to 2 years
Measure: Number; unit: Participants
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Participants
  Subjects with Grade 3 abnormality | 5
  Subjects with Grade 4 abnormality | 5
  Subjects with Grade 5 abnormality | 0

14. Secondary Outcome: Number of Abnormalities (Grade ≥3) in Laboratory Test Values
Description: Abnormalities in laboratory test values in overall study period were analyzed. Severity of abnormalities were evaluated using CTCAE.
Time Frame: Up to 2 years
Measure: Number; unit: Events
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
Events
  Grade 3 abnormalities | 33
  Grade 4 abnormalities | 39
  Grade 5 abnormalities | 0

15. Secondary Outcome: Pharmacokinetic Parameters (Cmax)
Description: Plasma pharmacokinetics (Cmax) of unchanged bendamustine
Time Frame: On Day 1 only
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
ng/mL | 8795.769 (3907.460)

16. Secondary Outcome: Pharmacokinetic Parameters (Tmax)
Description: Plasma pharmacokinetics (tmax) of unchanged bendamustine
Time Frame: On Day 1 only
Measure: Mean (Standard Deviation); unit: h
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
h | 1.00 (0.00)

17. Secondary Outcome: Pharmacokinetic Parameters (AUC)
Description: Plasma pharmacokinetics (AUC) of unchanged bendamustine
Time Frame: On Day 1 only
Measure: Mean (Standard Deviation); unit: ng・h/mL
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
ng・h/mL | 12315.992 (7900.579)

18. Secondary Outcome: Pharmacokinetic Parameters (t1/2)
Description: Plasma pharmacokinetics (t1/2) of unchanged bendamustine
Time Frame: On Day 1 only
Measure: Mean (Standard Deviation); unit: h
Arm/Group | SyB L-0501 + Prednisolone
Number analyzed (Participants) | 5
h | 0.44 (0.152)

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | SyB L-0501 + Prednisolone
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SyB L-0501 + Prednisolone (N=5)
Pneumonia (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Acute respiratory distress syndrome (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SyB L-0501 + Prednisolone (N=5)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Proctalgia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Malaise (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood albumin decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Blood potassium increased (Investigations) | 2
Blood sodium decreased (Investigations) | 1
Blood urea increased (Investigations) | 1
Blood uric acid decreased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
C-reactive protein increased (Investigations) | 3
CD4 lymphocytes decreased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 5
Neutrophil count increased (Investigations) | 3
Platelet count decreased (Investigations) | 5
Protein total decreased (Investigations) | 1
Weight increased (Investigations) | 2
White blood cell count decreased (Investigations) | 5
White blood cell count increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Scab (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Circulatory collapse (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No